CLINICAL TRIAL: NCT03305029
Title: Open-Label, Single-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of SCNT-hES-RPE Cells in Patients With Advanced Dry AMD
Brief Title: The Safety and Tolerability of Sub-retinal Transplantation of SCNT-hES-RPE Cells in Patients With Advanced Dry AMD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Won Kyung, Song, Principal Investigator, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA2015-08-141
Record Dates: First submitted 2016-07-06; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Dry Age Related Macular Degeneration
Keywords: Age related macular degeneration; embryonic stem cells; somatic cell nuclear transfer
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCNT-hES-RPE Cells (Experimental): Pars plana vitrectomy and Sub-retinal Transplantation of Human Somatic cell nuclear transfer Embryonic Stem Cell Derived Retinal Pigmented Epithelial Cells (SCNT-hES-RPE Cells) in Patients with Advanced Dry Age-related Macular Degeneration(AMD)
  Interventions: Drug: SCNT-hES-RPE Cells

INTERVENTIONS:
Drug: SCNT-hES-RPE Cells — Pars Plana Vitrectomy and Sub-retinal Transplantation of Human Somatic cell nuclear transfer Embryonic Stem Cell Derived Retinal Pigmented Epithelial(SCNT-hES-RPE) Cells in Patients with Advanced Dry Age-related Macular Degeneration

SUMMARY:
To evaluate the safety and tolerability of human somatic cell nuclear transfer embryonic stem cell derived retinal pigmented epithelial(SCNT-hES-RPE) cellular therapy in patients with advanced dry AMD

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of the SCNT-hES-RPEs, to assess the number of SCNT-hES-RPE cells to be transplanted in future studies and to evaluate on an exploratory basis potential efficacy endpoints to be used in future studies of SCNT-hES-RPE cellular therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female over 50 years of age.
2. Patient should be in sufficiently good health to reasonably expect survival for at least four years after treatment
3. Clinical findings consistent with advanced dry AMD with evidence of one or more areas of >250 microns of geographic atrophy (as defined in the Age-Related eye Disease Study [AREDS] study) involving the central fovea.
4. GA defined as attenuation or loss of RPE as observed by biomicroscopy, OCT, and FA.
5. The visual acuity (BCVA) of the eye to receive the transplant will be no better than 20/200 in Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity.
6. The visual acuity (BCVA) of the eye that is NOT to receive the transplant will be same or better than the eye to receive the transplant
7. Medically suitable to undergo vitrectomy and subretinal injection.
8. Medically suitable for general anesthesia or waking sedation, if needed.
9. If female and of childbearing potential, willing to medically acceptable methods of contraception during the study.
10. If male, willing to use barrier and spermicidal contraception during the study.
11. Willing to defer all future blood, blood component or tissue donation.
12. Able to understand and willing to sign the informed consent.

Exclusion Criteria:

1. Presence of active or inactive CNV in the eye to be treated.
2. Presence or history of retinal dystrophy, retinitis pigmentosa, chorioretinitis, central serious choroidopathy, diabetic retinopathy, other retinal vascular or degenerative disease other than ARMD, optic neuropathy, uveitis, intraocular inflammatory disease, retinal detachment repair or any other sight-threatening ocular disease.
3. Presence of glaucomatous optic neuropathy in the study eye, uncontrolled IOP, or use of two or more agents to control IOP (acetazolamide, beta blocker, alpha-1-agonist, prostaglandins, anhydrous carbonic inhibitors)
4. Cataract of sufficient severity likely to necessitate surgical extraction within 1 year.
5. Axial myopia of greater than -8 diopters.
6. Axial length greater than 28 mm.
7. Presence of significant lens opacities or other media opacity.
8. History of ocular lens removal within previous 3 months in the study eye.
9. History of ocular surgery in the study eye in the previous 3 months in the study eye.
10. History of malignancy or evidence of malignancy in screening test.
11. Medically not suitable for transplantation of an embryonic stem cell line: Any laboratory value which falls slightly outside of the normal range will be reviewed by the Medical Monitor and Investigators to determine its clinical significance. If it is determined not to be clinically significant, the patient may be enrolled into the study.

    * History of drug abuse, identified in medical history taking.
    * Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV.
    * Any immunodeficiency.
    * Negative cancer screening within previous 12 months: complete history & physical examination; negative chest roentgenogram (CXR); negative blood test(including CBC & manual differential); negative urinalysis (U/A); normal thyroid exam(T3, T4, TSH); if male, negative for prostate specific antigen (PSA); negative for upper gastrointestinal series or esophagogastroduodenoscopy; negative for α-fetoprotein(AFP); negative fecal occult blood test & negative colonoscopy; if female, normal clinical breast exam and, negative mammogram, negative breast ultrasonography; if female, normal pelvic examination with Papanicolaou smear;
    * Any of the below criteria of diabetes : Fasting blood glucose≥126mg/dl; random plasma glucose with typical symptoms of diabetes≥200mg/dl; HbA1c ≥ 7%
12. History of myocardial infarction or cerebrovascular accident in previous 12 months.
13. History of cognitive impairments or dementia which may impact the patients ability participate in the informed consent process and to appropriately complete evaluations.
14. Current participation in any other clinical trial.
15. Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.
16. If female, pregnancy or lactation.
17. Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Safety of SCNT-hES-RPE cells | 60 months
  The transplantation of SCNT-hES-RPE cells will be considered safe in the absence of:
  1. Any grade 2 (NCI CTCAE V4.03) or greater adverse event related to the cell product
  2. Any evidence that the cells are contaminated with an infectious agent
  3. Any evidence that the cells show tumorigenic potential

SECONDARY OUTCOMES:
● Change in the mean of BCVA | 60 months
  Best corrected ETDRS visual acuity scores
● Autofluorescence photography | 60 months
  Autofluorescence photography of GA
● Reading speed | 60 months
  MNReading speed measurements
● Structural evidence (OCT imaging, fluorescein angiography, autofluorescense photography, slitlamp examination with fundus phot ography) that cells have been implanted in the correct location | 60 months
  Evidence of structural changes

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No